CLINICAL TRIAL: NCT02980211
Title: Clinical, Radiographic and Histologic Evaluation of a Novel Alveolar Ridge Reconstruction Approach in Post-Extraction Dehiscence Defects: A Case Series Study
Brief Title: Treatment of Post-Extraction Dehisced Socket - A Case Series Study
Acronym: OSTEO2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gustavo Avila-Ortiz DDS, MS, PhD (Other)
Collaborators: Osteogenics Biomedical (Industry)
Responsible Party: Sponsor-Investigator, Gustavo Avila-Ortiz DDS, MS, PhD, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201612718
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Tooth Loss
Keywords: Alveolar Bone; Alveolar Ridge; Bone Resorption; Bone Grafting; Barrier Membrane
MeSH Terms: conditions — Tooth Loss; Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tooth Extraction and Graft Dehisced Socket (Experimental): Treatment of dehiscence defects at the time of tooth extraction using a minimally-invasive GBR technique that involves the application of a particulate bone allograft and a non-resorbable PTFE membrane.
  Interventions: Drug: Alveolar Ridge Reconstruction

INTERVENTIONS:
Drug: Alveolar Ridge Reconstruction — Reconstruction of dehiscence defects in extraction sockets with a minimally invasive technique using a particulate bone allograft and a non-absorbable dense polytetrafluoroethylene (dPTFE) membrane

SUMMARY:
PURPOSE The purpose of this case series is to clinically, radiographically and histologically evaluate the treatment of dehiscence defects in extraction sockets using a minimally-invasive GBR technique that involves the application of a particulate bone allograft and a non-resorbable PTFE membrane.

METHODS Subjects with single-rooted teeth indicated for extraction and interested in future implant therapy for tooth replacement will be recruited on the basis of an eligibility criteria. A buccal or lingual dehiscence defect must strongly be suspected or confirmed upon clinical examination in order for the subject to qualify for study inclusion. A cone-beam computer tomography (CBCT) scan of the arch containing the tooth to be extracted will be obtained prior to tooth extraction. Following minimally invasive tooth extraction and debridement, the socket will be evaluated to verify the presence of a dehiscence defect affecting at least 50% of the bony plate height. After creating a soft tissue 'pouch' using tunneling instruments, a non-absorbable dense-PTFE (dPTFE) barrier membrane that will be trimmed to a size and shape that would allow for complete extension over the existing defect will be tucked between the mucosa and the alveolar bone. Then, the extraction socket will be grafted with particulate allograft and the access to the socket will be sealed with an extension of the membrane and an external cross mattress suture. Subjects will be recalled at 1, 2 and 5 weeks to monitor healing and assess the level of discomfort using a visual analog scale at the end of each visit. At the 5-week visit, the membrane will be gently removed and the exposed area will be left to heal by secondary intention. At 20 weeks after tooth extraction a second CBCT will be obtained to radiographically evaluate the site for implant placement. Bone volumetric reconstructions of the alveolar ridge at baseline and at 20 weeks will be made using the CBCT data to assess changes affecting the bone housing. If the site has healed adequately, implant placement will be planned at 24 weeks after tooth extraction. A bone core biopsy will be obtained at the time of implant placement in order to histologically analyze the characteristics of the grafted substrate. Upon implant placement with primary stability a healing abutment will be placed and sutures will be given to achieve primary wound closure, as necessary. Subjects will return for the final study visit at 2 weeks following implant placement to evaluate the healing prior to being referred back to the restorative dentist.

DETAILED DESCRIPTION:
Visit 1 - Screening visit After reading and signing this informed consent form, you will complete a detailed medical and dental history form. We will review this form with you to ensure you can safely participate in the study. You will also have an oral exam to determine if you qualify for the study. If you are a woman of childbearing age, you will be tested for pregnancy. If you are pregnant or trying to become pregnant, you cannot participate in the study. You will also have one digital dental x-ray of the area for tooth extraction, if not available already, which is standard of care. You will also have dental impressions (molds of your teeth), which are made in a non-invasive manner to collect data for some of the research measurements. This visit will last between 1 and 1.5 hours.

Visit 2 - Baseline visit In less than 10 weeks after the screening visit, you will have the tooth extraction and bone grafting, which will be just like the procedure performed for patients who are not enrolled in the study and present a similar clinical scenario. Before the surgical procedure, a special dental x-ray scan known as cone beam computed tomography (CBCT) will be taken for the purpose of collecting research measurements. The CBCT scan generates 3D images of your teeth and surrounding tissues. After numbing the area, clinical measurements will be gathered. These measurements are non-invasive (do not involve cutting your body or putting instruments inside it) and will not harm the gums or surrounding teeth. The extraction (removal of the tooth) will be performed and the tooth socket (the area surrounding the tooth that was removed) will be cleaned, which is what would happen to patients who are not enrolled in the study. At this time, additional measurements of the area will be taken. These measurements will not cause you any extra discomfort, since that area will be numbed. Then, the socket grafting technique will be performed. The treatment will consist on the combination of a bone grafting material from a human donor (EnCore, Osteogenics Biomedical Inc.) and a non-dissolvable barrier membrane (Cytoplast TXT-200, Osteogenics Biomedical Inc.), to protect the bone graft and that will be removed in 5 weeks. You will be given prescriptions for an antibiotic, a pain reliever and a mouth rinse. You will also receive home care instructions before you leave. This visit will last about between 1.5 to 2 hours.

Visits 3, 4, 5 and 6 - Post-operative follow up visits You will return to the clinic at 1, 2, 5 and 20 weeks, which is standard of care in many cases of tooth extraction and grafting. In these visits, you will have an oral exam, check-up, and the researchers will monitor how well you are healing. These visits will last approximately 30 minutes.

At the 5-week visit, the barrier membrane will be removed. You will not have to be numbed for this.

Additionally, only at the 20-week visit after tooth extraction, a second CBCT x-ray scan will be obtained to determine how much bone is available after the healing period to plan the implant placement and for research measurements. The second CBCT x-ray scan will allow your surgical doctor to evaluate the amount of bone volume and is standard of care when planning for dental implant placement. A dental impression (mold) will be made to collect information about the gum tissue. Recommendations on further treatment, including the potential for implant therapy or possible additional grafting, will be provided based on the findings from this visit.

Visit 7 - Implant placement visit If you can receive the implant, a surgical placement visit will be scheduled at approximately 24 weeks after tooth extraction. After numbing the area, a small gum flap will be opened to access the area underneath that was bone grafted. A bone sample biopsy will be taken and analyzed for research purposes. This bone would be disposed otherwise, since a bed must be created in the bone to allow for implant placement. After an adequate space for implant placement is created in your bone, the implant will be placed. If implant primary stability (sufficient retention) is not achieved, the doctor may need to place a larger implant (in length, diameter or both) or, if this is not possible, discontinue the procedure and plan for delayed implant placement at another time. If this is the case, the study will cover the costs associated with additional grafting and implant placement. Upon implant placement, your gums will be stitched and you will be given prescriptions for an antibiotic, a pain reliever and a mouth rinse. You will also receive home care instructions before you leave. This visit will last between 1.5 and 2 hours.

Visit 8 - Post-operative follow up visit You will be seen by your surgical doctor for a postoperative visit at approximately 2 weeks after the implant is placed to monitor the healing and to remove sutures, which is standard of care. You will have an oral exam, check-up, and the researchers will monitor how well you are healing. These visits will last approximately 30 minutes. This is the last visit of the study.

ELIGIBILITY:
INCLUSION CRITERIA

* Provision of informed consent
* Age: 18 years or older
* Subjects with a single-rooted tooth indicated for extraction bounded by stable, natural teeth
* Tooth planned for extraction must have a dehiscence defect in the surrounding bone, observed clinically and/or radiographically, that affects at least 50% of the bone height
* Subjects must be interested in replacing the tooth with a single implant-supported fixed restoration
* Subjects must be able and willing to follow instructions related to the study procedures
* Subjects must have read, understood and signed an informed consent form

EXCLUSION CRITERIA

* Mandibular incisors
* Subjects with a history of organ failure (e.g. liver, kidney)
* Subjects with severe hematologic disorders, such as hemophilia or leukemia
* Subjects with uncontrolled and/or severe metabolic bone diseases or disorders, such as osteoporosis, thyroid disorders or Paget's disease
* Subjects taking any medication or supplement known to largely influence bone metabolism, such as IV bisphosphonates, long-term history of oral bisphosphonates or chronic intake of glucocorticoids
* Pregnant women (as indicated by positive serum HCG test) or nursing mothers
* Subjects with conditions that would result in compromised healing (e.g. poorly controlled diabetes, active heavy tobacco use [>10 cigs/day])
* Subjects who, at the discretion of the investigators, would be unsuitable candidates for the study due to safety, psychological or practical reasons (e.g. known allergies to any product used for the study, limited mouth opening, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Avila-Ortiz, DDS, MS, PhD, Principal Investigator — College of Dentistry
Locations (1):
- University of Iowa College of Dentistry - Craniofacial Clinical Research Program, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tooth Extraction and Graft Dehisced Socket
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tooth Extraction and Graft Dehisced Socket
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.82 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Bone Volumetric Reduction From Baseline to 20 Weeks Post-extraction
Description: Alveolar bone volumetric reduction from baseline to 20 weeks using CBCT scans
Time Frame: Baseline and 20 weeks post-extraction
Population: Two of the 17 DICOM datasets could not be analyzed due to extensive scattering, therefore the final sample size for this outcome was 15
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Tooth Extraction and Graft Dehisced Socket
Number analyzed (Participants) | 15
mm3 | 73.26 (77.27)

ADVERSE EVENTS:
Time Frame: 24 weeks post-extraction
Arm/Group | Tooth Extraction and Graft Dehisced Socket
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tooth Extraction and Graft Dehisced Socket (N=17)
Premature barrier membrane exfoliation (Surgical and medical procedures) | 1 (1) — One patient decided to remove the membrane himself between 2 and 5 weeks because it was "bothersome"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT02980211/Prot_SAP_000.pdf